CLINICAL TRIAL: NCT00056212
Title: Evaluating Yoga for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001215-01 (NIH)
Record Dates: First submitted 2003-03-07; First posted 2003-03-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Yoga; Exercise

INTERVENTIONS:
Behavioral: Yoga
Behavioral: Exercise

SUMMARY:
This study will compare the effectiveness of yoga classes, exercise classes, and a self-care book in the management of pain and function for people with low back pain.

DETAILED DESCRIPTION:
Back problems are among the most prevalent conditions affecting adults and are a leading reason for using complementary or alternative medical (CAM) therapies. Despite the common use of CAM therapies for back pain, little is known about how they compare with conventional treatments. This study will lay the groundwork for a full-scale trial that compares yoga with conventional exercise and usual care for chronic low back pain.

This study will randomize 30 people with chronic low back pain to each of the following groups: yoga, a conventional therapeutic exercise program, and usual care. There will be 12 weeks of weekly treatment and follow-up assessments via phone at 6, 12, and 26 weeks to measure each treatment's impact on symptoms, function, quality of life, and utilization and costs of back pain related care.

ELIGIBILITY:
Inclusion criteria:

* Group Health Cooperative enrollee
* Uncomplicated low back pain
* At least moderate pain levels

Exclusion criteria:

* Sciatica persisting 3 or more months after physician visit
* History of cancer (other than nonmelanoma skin cancer)
* Severe disk problems
* Unstable medical conditions
* Back surgery within past 3 years
* Physically unable to do the yoga or exercise classes and homework
* Unable to attend classes
* Currently doing yoga
* Taken exercise class for back pain within past year
* Currently in litigation for back pain
* Seeking other treatment for back pain

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2002-07; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Sherman, Ph.D., Principal Investigator — Center for Health Studies, Group Health Cooperative
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Result] Sherman KJ, Cherkin DC, Erro J, Miglioretti DL, Deyo RA. Comparing yoga, exercise, and a self-care book for chronic low back pain: a randomized, controlled trial. Ann Intern Med. 2005 Dec 20;143(12):849-56. doi: 10.7326/0003-4819-143-12-200512200-00003. PMID 16365466